CLINICAL TRIAL: NCT06626243
Title: An International Multicenter Retrospective Analysis of RATS, VATS and Open Lung Resections After Neoadjuvant Chemo-immunotherapy
Brief Title: Analysis of RATS, VATS and Open Lung Resections After Neoadjuvant Chemo-immunotherapy in Patients Performed in Five Referred Centers
Acronym: IMMUNORATS
Status: Recruiting | Type: Observational
Sponsor: Scientific Institute San Raffaele (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); Istituto Clinico Humanitas (Other); Regina Elena Cancer Institute (Other); Baptist Health South Florida (Other); West Virginia University (Other)
Responsible Party: Principal Investigator, Pierluigi Novellis, Principal Investigator, Scientific Institute San Raffaele
Other Study IDs: CET 380-2024
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Video-Assisted Thoracoscopic Surgery; Robot-Assisted Thoracoscopic Surgery; open approach
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Robotic Approach: Adult patients diagnosed with locally advanced and resectable non-small cell lung cancer (NSCLC) who underwent robotic lung resection
- video-assisted thoracoscopic surgery (VATS) Approach: Adult patients diagnosed with locally advanced and resectable non-small cell lung cancer (NSCLC) who underwent video-assisted thoracoscopic surgery (VATS) lung resection
- Open Approach: Adult patients diagnosed with locally advanced and resectable non-small cell lung cancer (NSCLC) who underwent open lung resection

SUMMARY:
The study is a retrospective observational study. The study is designed to be multicentric and international and it will analyze medical records from selected patients diagnosed with locally advanced and resectable NSCLC who underwent lung resection by robotic, VATS and open approach after receiving neoadjuvant chemo-immunotherapy.

There are no risks for the patients, as this is a retrospective data collection.

DETAILED DESCRIPTION:
The use of neoadjuvant chemo-immunotherapy for the treatment of non-small cell lung cancer (NSCLC) is increasing. However, there is limited research comparing the feasibility and oncologic efficacy of robot-assisted thoracoscopic surgery (RATS), video-assisted thoracoscopic surgery (VATS), and open lung resection, in patients already treated with neoadjuvant chemo-immunotherapy. This study aims to evaluate the benefits of RATS compared to VATS and open surgery in terms of short-term outcomes for patients with NSCLC undergoing neoadjuvant chemo-immunotherapy.

All adult patients diagnosed with locally advanced and resectable NSCLC who underwent lung resection from 01-01-2016 to 31-03-2024 by robotic, VATS and open approach after receiving neoadjuvant chemo-immunotherapy will be included.

Patients are divided into three groups: robotic lung resection; video-assisted thoracoscopic (VATS) lung resection; open lung resection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinical or pathological stage IIB (T1-2, hilar N1, M0) and III (any T, N1-2, M0) NSCLC surgically treated with robotic, VATS and open approach with radical intent from 1st of January 2016 to 31st of March 2024
* Received neoadjuvant chemo-immunotherapy or immunotherapy alone
* Age >= 18 years old at the moment of surgery

Exclusion Criteria:

* Age <18 years old at the moment of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed locally advanced and resectable non-small cell lung cancer (NSCLC) who underwent lung resection from 01-01-2016 to 31-03-2024 by robotic, video-assisted thoracoscopic (VATS), and open approaches after receiving neoadjuvant chemo-immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
The perioperative complication of video-assisted thoracoscopic surgery (VATS) approach | 30-90 days after surgery
  The investigators will measure the perioperative complications of VATS approach in patients who received neoadjuvant chemo-immunotherapy. Complications will be categorized according to the Clavien-Dindo scale.
The perioperative complications of robotic approach | from the surgery at 30-90 days after
  The investigators will measure the perioperative complications of robotic lung resection in patients who received neoadjuvant chemo-immunotherapy. Complications will be categorized according to the Clavien-Dindo scale.
The perioperative complications of the open approach | 30-90 days after surgery
  The investigators will measure the perioperative complications of open approach in patients who received neoadjuvant chemo-immunotherapy. Complications will be categorized according to the Clavien-Dindo scale.

SECONDARY OUTCOMES:
Duration of surgery | from 30 days after surgery
  Duration of the surgery based on the approach measured in minutes
Quality of lymphadenectomy | from 30 days after surgery
  Number of lymphonodes station resected
Conversion rate | from 30 days after surgery
  Number of surgery procedures converted
Radicality of the resection | from 30 days after surgery
  Radicality of the resection in the approaches
Oncological treatment | from 30 days after surgery
  Response of the patient to oncological treatment
Survival analysis | from 3 to 5 years after surgery
  Presence or absence of local and distant relapse

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Baptist Health South Florida, Miami, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - West Virginia University, Morgantown, West Virginia
- Italy (3):
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Scientific Institute Ospedale San Raffaele, Milan
  - Regina Elena National Cancer Institute, Rome